CLINICAL TRIAL: NCT01709929
Title: A Multicentre, Open Label, Nonrandomised, Safety Study in Subjects Using Insulin Detemir for the Treatment of Insulin Dependent Type 1 or Type 2 Diabetes Mellitus
Brief Title: Safety of Insulin Detemir for the Treatment of Insulin Dependent Type 1 or Type 2 Diabetes Mellitus
Acronym: PREDICTIVE™
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN304-1713
Record Dates: First submitted 2012-10-16; First posted 2012-10-18 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Insulin detemir (Experimental)
  Interventions: Drug: insulin detemir

INTERVENTIONS:
Drug: insulin detemir — Administered subcutaneously (s.c., under the skin). Dose individually adjusted.

SUMMARY:
This trial is conducted in North America. The aim of this trial is to evaluate the safety of insulin detemir for the treatment of diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 1 or type 2 diabetes
* Using a basal/bolus insulin regimen

Exclusion Criteria:

* Subjects who are unlikely to comply with protocol, e.g., uncooperative attitude, inability to return for the final visit
* Subjects who previously enrolled in this study
* Subjects with a hypersensitivity to insulin detemir or to any of the excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2287 (Actual)
Dates: Start 2005-10; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Incidence of serious adverse drug reactions (SADRs) including major hypoglycaemic events

SECONDARY OUTCOMES:
Number of adverse events (all and serious)
Number of all hypoglycaemic events
Change in weight
HbA1c (glycosylated haemoglobin)
Treatment satisfaction as assessed by Insulin Treatment Satisfaction Questionnaire (ITSQ-22)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Mississauga, Canada

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com